CLINICAL TRIAL: NCT00265798
Title: A Phase 2 Study of BAY 43-9006 for Imatinib- and Sunitinib Resistant Gastrointestinal Stromal Tumor
Brief Title: Sorafenib in Treating Patients With Malignant Gastrointestinal Stromal Tumor That Progressed During or After Previous Treatment With Imatinib Mesylate and Sunitinib Malate
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00116; NCI-2009-00116 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-7028; CDR0000739566; 13780A (Other: University of Chicago Comprehensive Cancer Center); 7028 (Other: CTEP); N01CM62201 (NIH); N01CM62206 (NIH); N01CM62207 (NIH); N01CM62209 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Results first posted 2014-01-21 (Estimated); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sorafenib Tosylate

INTERVENTIONS:
Drug: Sorafenib Tosylate
  Other Names: BAY 43-9006 Tosylate; BAY 54 9085; BAY 54-9085; BAY 549085; BAY-54-9085; BAY549085; Nexavar; sorafenib

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with malignant gastrointestinal stromal tumor that progressed during or after previous treatment with imatinib mesylate and sunitinib malate. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate of patients with imatinib and sunitinib-resistant malignant gastrointestinal stromal tumor who are treated with BAY 43-9006.

SECONDARY OBJECTIVES:

I. To determine the toxicity experienced by patients with imatinib and sunitinib -resistant malignant gastrointestinal stromal tumor who are treated with BAY 43-9006.

II. To determine progression-free survival and overall survival in patients with imatinib and sunitinib -resistant malignant gastrointestinal stromal tumor who are treated with BAY 43-9006.

TERTIARY OBJECTIVES:

I. To examine if mutational status of KIT and PDGFA in patients with imatinib- and sunitinib resistant malignant gastrointestinal stromal tumor correlate with response to BAY 43-9006.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior treatment with imatinib mesylate and sunitinib malate (imatinib mesylate- and sunitinib malate-responsive disease vs primary imatinib mesylate- and sunitinib malate-refractory disease).

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastrointestinal stromal tumor

  * Not amenable to curative surgery
* Kit-expressing tumor
* Disease progression (i.e., new lesion or 20% increase in unidimensional tumor size) on or after treatment with imatinib mesylate and sunitinib malate
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques OR > 10 mm by spiral CT scan

  * Only site of measurable disease must be outside of previously irradiated area
* No known brain metastases
* Performance status - ECOG 0-2
* More than 3 months
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin normal
* AST and ALT < 2.5 times upper limit of normal
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance > 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to sorafenib
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No evidence of bowel perforation or obstruction
* No prior angiogenesis inhibitors
* No immunotherapy after the last dose of imatinib mesylate or sunitinib malate
* No chemotherapy or chemoembolization therapy after the last dose of imatinib mesylate or sunitinib malate
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* At least 14 days since prior imatinib mesylate or sunitinib malate
* No prior sorafenib
* No prior inhibitors of MAPK-signaling intermediates
* No other investigational agent after the last dose of imatinib mesylate or sunitinib malate
* Concurrent anticoagulation therapy with warfarin allowed provided the following criteria are met:

  * On a therapeutic stable warfarin dose
  * INR ≤3
  * No active bleeding or pathologic condition that confers a high risk of bleeding
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent administration of any of the following:

  * Enzyme-inducing antiepileptic drugs (e.g., carbamazepine, phenytoin, or phenobarbital)
  * Hypericum perforatum (St. John's wort)
  * Rifampin
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-09-14 (Actual); Primary Completion 2010-02-11 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (6):
- United States (6):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 6 centers between 2006 and 2009
Groups:
- Sorafenib: Patients receive oral Sorafenib 400mg twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sorafenib
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 38
Study Cohort [Number; unit: participants] — Participants were classified as having either imatinib-resistant disease or imatinib- and sunitinib-resistant disease
  participants
    Imatinib-resistant | 6
    Imatinib- and sunitinib-resistant | 32
Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status scores on a scale of 0-5, higher is worse 0= Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light/sedentary nature
  2. Ambulatory and capable of all selfcare, unable to carry out any work activities. Up and about > 50% of waking hours
  3. Capable of only limited selfcare, confined to bed/chair > 50% of waking hours
  4. Completely disabled. Cannot carry on any selfcare. Totally confined to bed/chair
  5. Dead
  participants
    0 | 18
    1 | 18
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response (complete response (CR)+ partial response (PR)) will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR is the disappearance of all target lesions. PR requires at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Computed Tomography (CT) scans for disease reassessment will be obtained pre-therapy and every 8 weeks. In addition to a baseline scan, confirmatory scans will also be obtained 4 weeks following initial documentation of objective response.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | Sorafenib
Number analyzed (Participants) | 38
percentage of partcipants | 13 [4 to 28]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be defined as time from the start of treatment until progression (documented according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions) or death, whichever comes first.
  CT scans for disease reassessment will be obtained pre-therapy and every 8 weeks.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 38
months | 5.2 [3.4 to 7.4]

3. Secondary Outcome: Overall Survival
Description: Overall survival will be defined as time from the start of treatment until death from any cause.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib
Number analyzed (Participants) | 38
months | 11.6 [8.8 to 14.3]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of treatment
Description: Adverse events of grade 3 or higher at least possibly related to treatment are reported
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 5/38
Other Adverse Events (participants affected / at risk) | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=38)
Thrombosis (Vascular disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=38)
Diarrhea (Gastrointestinal disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 2
Hypertension (Vascular disorders) | 7
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less